CLINICAL TRIAL: NCT01228123
Title: Prospective Randomised Clinical Trial of the Effect of Continuous Versus Intermittent Renal Replacement Therapy on the Mortality and Outcome of Acute Renal Failure in ICU Patients
Brief Title: Clinical Trial Comparing Continuous Versus Intermittent Hemodialysis in ICU Patients
Acronym: CONVINT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: investigator initiated trial (see adress below), Charite University Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CONVINT
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2010-07

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVVH arm (Active Comparator)
  Interventions: Other: RRT for acute kidney failure using the CVVH method
- IHD arm (Active Comparator)
  Interventions: Other: RRT for acute kidney failure using the IHD (intermittent HD)

INTERVENTIONS:
Other: RRT for acute kidney failure using the CVVH method — patients randomized to receive CVVH
  Other Names: does not apply
  Arms: CVVH arm
Other: RRT for acute kidney failure using the IHD (intermittent HD) — patients randomized to receive IHD
  Other Names: does not apply
  Arms: IHD arm

SUMMARY:
The mortality of acute renal failure (ARF) remains to be high (around 60-70%) despite manifold improvements in ICU care. At present, it is not clear if the method chosen for renal replacement therapy, i.e. intermittent haemodialysis (IHD) or continuous haemofiltration (CVVH), might impact on the outcome of these patients. For this purpose, a prospective randomised clinical study of the effect of continuous versus intermittent renal replacement therapy on the mortality and outcome of acute renal failure will be performed.

DETAILED DESCRIPTION:
please see above

ELIGIBILITY:
Inclusion Criteria:

* all ICU patients requiring renal replacement therapy

Exclusion Criteria:

* patient denies informed consent
* patient not requiring intensive care therapy
* kidney transplanted patients
* chronic renal failure (serum creatinine > 3mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2002-01; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Survival at 2 weeks after RRT | 2 weeks after RRT in follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Achim Joerres, MD, Principal Investigator — Charite University Medicine
Locations (1):
- Charite University Medicine, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356
- [Derived] Schefold JC, von Haehling S, Pschowski R, Bender T, Berkmann C, Briegel S, Hasper D, Jorres A. The effect of continuous versus intermittent renal replacement therapy on the outcome of critically ill patients with acute renal failure (CONVINT): a prospective randomized controlled trial. Crit Care. 2014 Jan 10;18(1):R11. doi: 10.1186/cc13188. PMID 24405734